CLINICAL TRIAL: NCT01660035
Title: The REsynchronization reVErses Remodeling in Systolic Left vEntricular Dysfunction (REVERSE) Post Approval Study
Brief Title: The Product Surveillance Registry REVERSE Post Approval Study
Acronym: PSR-REVERSE
Status: Completed | Type: Observational
Sponsor: Medtronic (Industry)
Responsible Party: Sponsor
Other Study IDs: PSR-REVERSE
Record Dates: First submitted 2012-08-06; First posted 2012-08-08 (Estimated); Last update posted 2022-04-18 (Actual); Status verified 2022-04

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of the REVERSE Post Approval Study (PAS) is to confirm the benefit observed in the REVERSE and RAFT pivotal studies in "real-world" clinical practice.

DETAILED DESCRIPTION:
The REVERSE PAS will estimate the 3-year survival probability of freedom from heart failure hospitalization and heart failure events in patients implanted with a Medtronic CRT-D device who meet the expanded indication criteria with a QRS duration ≤ 150 ms.

ELIGIBILITY:
Inclusion Criteria:

* Patient or legally authorized representative provides written authorization and/or consent per institution and geographical requirements
* Patient has or is intended to receive or be treated with a Medtronic CRT-D who meets the expanded CRT-D indication criteria with a QRS ≤ 150ms
* Patient within 30 days of implant

Exclusion Criteria:

* Patient who is, or will be, inaccessible for follow-up
* Patient with exclusion criteria required by local law
* Patient is currently enrolled in or plans to enroll in any concurrent drug and/or device study that may confound results

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Heart failure patients that are implanted with a Medtronic CRT-D device and meet the expanded indication criteria.
Sampling Method: Non-Probability Sample
Enrollment: 155 (Actual)
Dates: Start 2012-04 (Actual); Primary Completion 2022-04 (Actual); Study Completion 2022-04 (Actual)

PRIMARY OUTCOMES:
Survival from Heart Failure Hospitalization and All-Cause Mortality | 3 years
  To estimate the 3-year survival probability of freedom from heart failure hospitalization or all-cause death for patients implanted with a Medtronic CRT-D device meeting the approved expanded indication criteria with a QRS duration ≤ 150ms.
Survival from Heart Failure Event and All-Cause Mortality | 3 years
  To estimate the 3-year survival probability of freedom from heart failure event or all- cause death for patients implanted with a Medtronic CRT-D device meeting the approved expanded indication criteria with a QRS duration ≤ 150ms.

CONTACTS AND LOCATIONS:
Locations (123):
- United States (102):
  - Birmingham, Alabama
  - Anchorage, Alaska
  - Chandler, Arizona
  - Gilbert, Arizona
  - Jonesboro, Arkansas
  - Little Rock, Arkansas
  - Bakersfield, California
  - Chula Vista, California
  - Los Angeles, California
  - Rancho Mirage, California
  - Redwood City, California
  - Salinas, California
  - San Diego, California
  - Stanford, California
  - Torrance, California
  - Van Nuys, California
  - Colorado Springs, Colorado
  - Lakewood, Colorado
  - New Haven, Connecticut
  - Washington D.C., District of Columbia
  - Bradenton, Florida
  - Clearwater, Florida
  - Jacksonville, Florida
  - Safety Harbor, Florida
  - Albany, Georgia
  - Atlanta, Georgia
  - Marietta, Georgia
  - Evansville, Indiana
  - West Des Moines, Iowa
  - Kansas City, Kansas
  - Edgewood, Kentucky
  - Lexington, Kentucky
  - Louisville, Kentucky
  - Baton Rouge, Louisiana
  - Hyattsville, Maryland
  - Salisbury, Maryland
  - Silver Spring, Maryland
  - Takoma Park, Maryland
  - Lansing, Michigan
  - Marquette, Michigan
  - Ypsilanti, Michigan
  - Coon Rapids, Minnesota
  - Minneapolis, Minnesota
  - Robbinsdale, Minnesota
  - Rochester, Minnesota
  - Saint Cloud, Minnesota
  - Saint Paul, Minnesota
  - Hattiesburg Clinic, Hattiesburg, Mississippi
  - Columbia, Missouri
  - Kansas City, Missouri
  - Lebanon, New Hampshire
  - Morristown, New Jersey
  - Ocean City, New Jersey
  - Ridgewood, New Jersey
  - Albuquerque, New Mexico
  - Bay Shore, New York
  - Huntington, New York
  - Manhasset, New York
  - New Hyde Park, New York
  - New York, New York
  - Poughkeepsie, New York
  - Staten Island, New York
  - The Bronx, New York
  - Utica, New York
  - Charlotte, North Carolina
  - Durham, North Carolina
  - Raleigh, North Carolina
  - Akron, Ohio
  - Cincinnati, Ohio
  - Cleveland, Ohio
  - Columbus, Ohio
  - Toledo, Ohio
  - Oklahoma City, Oklahoma
  - Portland, Oregon
  - Allentown, Pennsylvania
  - Bethlehem, Pennsylvania
  - Danville, Pennsylvania
  - Erie, Pennsylvania
  - Lancaster, Pennsylvania
  - Philadelphia, Pennsylvania
  - Pittsburgh, Pennsylvania
  - Wilkes-Barre, Pennsylvania
  - Wynnewood, Pennsylvania
  - Columbia, South Carolina
  - Germantown, Tennessee
  - Nashville, Tennessee
  - Austin, Texas
  - Dallas, Texas
  - Fort Worth, Texas
  - Houston, Texas
  - Plano, Texas
  - San Antonio, Texas
  - The Woodlands, Texas
  - Burlington, Vermont
  - Charlottesville, Virginia
  - Falls Church, Virginia
  - Leesburg, Virginia
  - Olympia, Washington
  - Spokane, Washington
  - Tacoma, Washington
  - Madison, Wisconsin
  - Milwaukee, Wisconsin
- Leuven, Belgium
- Canada (5):
  - Calgary, Alberta
  - London, Ontario
  - Ottawa, Ontario
  - Montreal, Quebec
  - Québec, Quebec
- France (2):
  - La Rochelle
  - Nantes
- Germany (4):
  - Essen
  - Hanover
  - Homburg
  - Ulm
- Reggio Emilia, Italy
- Netherlands (4):
  - Eindhoven
  - Maastricht
  - Nieuwegein
  - Rotterdam
- Skövde, Sweden
- Zurich, Switzerland
- United Kingdom (2):
  - Liverpool
  - Middlesbrough